CLINICAL TRIAL: NCT04854044
Title: Phase 1b Study of ONC201 and Radiotherapy in Preoperative Recurrent Glioblastoma (GBM) Patients
Brief Title: ONC201 and Radiation Therapy Before Surgery for the Treatment of Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The P.I. is not prepared to move forward at this thime
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oncoceutics, Inc. (Industry); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-000054; NCI-2021-02121 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-000054 (Other: UCLA / Jonsson Comprehensive Cancer Center); P50CA211015 (NIH)
Record Dates: First submitted 2021-03-31; First posted 2021-04-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-03

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliosarcoma; Recurrent Supratentorial Glioblastoma; Supratentorial Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — TIC10 compound; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ONC201, radiation therapy, resection) (Experimental): Patients undergo radiation therapy for 10 fractions over 2 weeks, and receive ONC201 PO daily on days 1, 2, 8, and 9. Beginning 24 hours after completion of radiation therapy, patients undergo surgical resection. Beginning 7 days from last pre-surgery dose of ONC201, patients receive ONC201 PO daily on two consecutive days weekly (2 days on/5 days off) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Radiation: Radiation Therapy; Procedure: Resection
- Arm II (ONC201, radiation therapy, resection) (Experimental): Patients undergo radiation therapy for 10 fractions over 2 weeks. Beginning 24 hours after completion of radiation therapy, patients undergo surgical resection. After recovery from surgery, patients receive ONC201 PO daily on two consecutive days weekly (2 days on/5 days off) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Radiation: Radiation Therapy; Procedure: Resection

INTERVENTIONS:
Drug: Akt/ERK Inhibitor ONC201 — Given orally
  Other Names: ONC201; TIC10
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase I trial studies the effects of ONC201 in combination with standard of care radiation therapy in treating patients with glioblastoma that has come back (recurrent). ONC201 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy photons to kill tumors cells and shrink tumors. Giving ONC201 in combination with radiation therapy may help treat patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of Akt/ERK Inhibitor ONC201 (ONC201) in combination with radiotherapy before a tumor resection in recurrent glioblastoma (GBM) patients.

II. To determine the ability of ONC201 to decrease glioblastoma-initiating cells as determined by percentage of neurosphere formation of treated brain tumor tissues compared to non-treated brain tumor tissues.

SECONDARY OBJECTIVES:

I. To determine the ability of ONC201 to decrease glioblastoma-initiating cells as determined by expression of glioma stem cells using ribonucleic acid-sequencing (RNA-Seq) of treated brain tumor tissues compared to non-treated brain tumor tissues.

II. To assess the ability of ONC201 to inhibit Akt by evaluating progressive disease (PD) markers by immunohistochemistry such as Sox2, Oct3/4, Nanog, Akt and p-Akt, GSK3 and pGSK3alpha.

EXPLORATORY OBJECTIVES:

I. To estimate progression-free survival (PFS) and overall survival (OS). II. To determine the immunogenicity of the combination of ONC201 + radiation therapy (RT) via immune cell studies.

III. To determine if the combination of ONC201 + RT leads to increase cholesterol synthesis.

IV. To determine molecular markers of response to ONC201 in correlation to survival such as DRD5 expression.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo radiation therapy for 10 fractions over 2 weeks, and receive ONC201 orally (PO) daily on days 1, 2, 8, and 9. Beginning 24 hours after completion of radiation therapy, patients undergo surgical resection. Beginning 7 days from last pre-surgery dose of ONC201, patients receive ONC201 PO daily on two consecutive days weekly (2 days on/5 days off) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo radiation therapy for 10 fractions over 2 weeks. Beginning 24 hours after completion of radiation therapy, patients undergo surgical resection. After recovery from surgery, patients receive ONC201 PO daily on two consecutive days weekly (2 days on/5 days off) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically proven glioblastoma or gliosarcoma which is progressive or recurrent following radiation therapy +/- chemotherapy
* Participants must have evaluable, supratentorial contrast-enhancing progressive or recurrent glioblastoma or gliosarcoma by magnetic resonance imaging (MRI) imaging within 14 days of study treatment initiation. Participants must be able to tolerate MRIs
* Participants can have any number of prior relapses
* Participants must have recovered from severe toxicity of prior therapy. The following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy or mitomycin C
  * 23 days from temozolomide chemotherapy
  * 4-weeks from other cytotoxic therapy unless noted above
  * 4 weeks or 5-half-lives (whichever is shorter) from any other investigational (not Food and Drug Administration [FDA]-approved) agents (including vaccines)
* Participants must be undergoing surgery that is clinically indicated as determined by their care providers. Patients must be eligible for surgical resection with the expectation that the surgeon is able to resect at least 300 mg of tumor with low risk of inducing neurological injury
* Participants must be undergoing radiotherapy that is clinically indicated as determined by their care providers. The field of radiation must overlap the area of tumor planned for surgical resection. Participants must have a minimum tumor size of 2 x 2 cm^2 based on MRI scan prior to surgery
* Participants must be 18 years of age or older
* Participants must have a Karnofsky performance status >= 60% (i.e. the participant must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 50 mL/min/1.73m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time/ partial thromboplastin time (APTT/PTT) =< 1.5 x institutional upper limit of normal (unless participant is receiving anticoagulant therapy as long as prothrombin time [PT] or aPTT is within therapeutic range of intended use of anticoagulants)
* Female participants of childbearing potential must have a negative urine or serum pregnancy test prior to study entry. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle stimulating hormone [FSH] levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Female participants of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 30 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 30 days after the last dose of study drug. Women who are nursing should discontinue nursing prior to starting study drug
* Participants must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with prior malignancies must be disease-free for >= three years
* Participants must be able to swallow whole capsules
* Participants must have at least 20 (preferably 40) slides of archival tumor tissue from a prior surgery demonstrating GBM
* Participants must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants receiving any other investigational agents or using an investigational device are ineligible
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 are ineligible
* Participants may not have had prior treatment with ONC201
* Participants may have had prior treatment with bevacizumab/VEGFR inhibitors, but last dose of treatment must be at least 4 weeks prior to the date of planned tumor resection
* Participants may not be on concurrent treatment with Optune device. Prior use of the device is allowable
* Participants must not have evidence of significant hematologic, renal, or hepatic dysfunction
* Participants with a history of any of the following within the last 6 months prior to study entry are ineligible:

  * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
  * Ischemic cerebrovascular event, including transient ischemic attack (TIA) and artery revascularization procedures
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
  * Placement of a pacemaker for control of rhythm
  * New York Heart Association (NYHA) class III or IV heart failure
* Participants with known significant active cardiovascular or pulmonary disease at the time of study entry are ineligible
* Participants receiving therapeutic agents known to prolong QT interval will be excluded. Patients on sertraline which has the conditional risk of prolonging the QT interval will be allowed on study if they hold sertraline on the day of ONC201 administration
* Participants using concomitant CYP3A4/5 inhibitors within 72 hours prior to starting study drug administration are ineligible
* Participants with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study because there is unknown risk of ONC201 on the fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother on ONC201, breastfeeding should be discontinued if the mother is treated with ONC201

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 90 days after the last study treatment
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Percentage of neurosphere formation | At the tumor resection during surgery
  A two-sample two-sided t-test will be performed to compare the percentage of neurosphere formation of treated brain tumor tissues and non-treated brain tumor tissues.

SECONDARY OUTCOMES:
Expression of glioma stem cells using ribonucleic acid-sequencing (RNA-Seq) | At the tumor resection during surgery
  Will be compared between treated brain tumor tissues and non-treated brian tumor tissues. Markers for expression of glioma stem cells as determined by RNA-Seq and makers indicating cellular pathways leading to formation of GICs, such as Sox2, Oct3/4, Nanog, Akt and p-Akt, GSK3 and pGSK3alpha, will be examined graphically and summarized by descriptive statistics. Changes in markers pre- and post- treatment will be assessed using paired t-tests or Wilcoxon signed rank test. Between-group differences in these markers will be assessed by two-sample t-test or Wilcoxon rank-sum test for quantitative variables and by Chi-squared test or Fisher's exact test for categorical ones.
Pharmacodynamic (PD) markers | At the tumor resection during surgery
  Evaluated by immunohistochemistry such as Sox2, Oct3/4, Nanog, Akt and p-Akt, GSK3 and pGSK3alpha. Markers for expression of glioma stem cells as determined by RNA-Seq and makers indicating cellular pathways leading to formation of GICs, such as Sox2, Oct3/4, Nanog, Akt and p-Akt, GSK3 and pGSK3alpha, will be examined graphically and summarized by descriptive statistics. Changes in markers pre- and post- treatment will be assessed using paired t-tests or Wilcoxon signed rank test. Between-group differences in these markers will be assessed by two-sample t-test or Wilcoxon rank-sum test for quantitative variables and by Chi-squared test or Fisher's exact test for categorical ones.

OTHER OUTCOMES:
Progression-free survival | Up to 4 years
  Kaplan-Meier (KM) curves and the median time to progression estimated from the KM curves will be provided for each group as appropriate. Log-rank test will be used to compare Group A versus Group B.
Overall survival | Up to 4 years
  KM curves and the median time to progression estimated from the KM curves will be provided for each group as appropriate. Log-rank test will be used to compare Group A versus Group B.
Pharmacodynamic markers | At the tumor resection during surgery
  Post-treatment tissues will be assessed for Pharmacodynamic markers (Sox2, Oct3/4, Nanog, Akt and p-Akt, GSK3 and pGSK3alpha) by RNA-seq and IHC to evaluate the immunogenicity of ONC201 for recurrent glioblastoma.
Determine if the combination of ONC201 + RT leads to increase cholesterol synthesis | At screening, pre-surgery, every 4 weeks post-surgery, and the end of study treatment, up to 48 months
  Cholesterol synthesis level will be evaluated via laboratory testing of RNA-seq.
Determine molecular markers of response to ONC201 in correlation to survival such as DRD5 expression | Up to 4 years
  Pre-treatment archival tumor tissue and post-treatment tumor tissue will be obtained to evaluate other molecular markers of response to ONC201 + RT, including pharmacodynamic markers such as DRD2 and DRD5.

CONTACTS AND LOCATIONS:
Overall Officials: Phioanh Nghiemphu, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States